CLINICAL TRIAL: NCT02887950
Title: Resistant Starch, Epigallocatechin Gallate and Chlorogenic Acid for Body Weight Loss in Overweight Menopausal Women: a Pragmatic, Randomised Clinical Trial.
Brief Title: Resistant Starch, Epigallocatechin Gallate and Chlorogenic Acid for Body Weight Loss in Menopause
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No benefit at iterim analysis
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Leonardo Medica Srl (Unknown)
Responsible Party: Principal Investigator, Riccardo Caccialanza, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20150021742
Record Dates: First submitted 2016-08-16; First posted 2016-09-02 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2019-02

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nutritional counseling (Active Comparator): Nutritional counseling consists in: personalized dietary prescription associated with dietetic advise (on a monthly basis and upon patient's request) by a registered dietician.
  Interventions: Other: Nutritional counseling
- Equikilon-3 months (Experimental): The patient will receive 2 sachets per day of a dietary supplement containing resistant starch, epigallocatechin gallate and chlorogenic acid (Equikilon) for 3 months and nutritional counseling.
  Nutritional counseling consists in: personalized dietary prescription associated with dietetic advise (on a monthly basis and upon patient's request) by a registered dietician.
  Interventions: Dietary Supplement: Equikilon-3 months
- Equikilon-6 months (Experimental): The patient will receive 2 sachets per day of a dietary supplement containing resistant starch, epigallocatechin gallate and chlorogenic acid (Equikilon) for 6 months and nutritional counseling.
  Nutritional counseling consists in: personalized dietary prescription associated with dietetic advise (on a monthly basis and upon patient's request) by a registered dietician.
  Interventions: Dietary Supplement: Equikilon-6 months

INTERVENTIONS:
Other: Nutritional counseling — Nutritional counseling consists in: personalized dietary prescription associated with dietetic advise (on a monthly basis and upon patient's request) by a registered dietician.
  Arms: Nutritional counseling
Dietary Supplement: Equikilon-3 months — The patient will receive 2 sachets per day of a dietary supplement containing resistant starch, epigallocatechin gallate and chlorogenic acid (Equikilon) for 3 months and nutritional counseling.
  Nutritional counseling consists in: personalized dietary prescription associated with dietetic advise (on a monthly basis and upon patient's request) by a registered dietician.
  Arms: Equikilon-3 months
Dietary Supplement: Equikilon-6 months — The patient will receive 2 sachets per day of a dietary supplement containing resistant starch, epigallocatechin gallate and chlorogenic acid (Equikilon) for 6 months and nutritional counseling.
  Nutritional counseling consists in: personalized dietary prescription associated with dietetic advise (on a monthly basis and upon patient's request) by a registered dietician.
  Arms: Equikilon-6 months

SUMMARY:
For women aged between 55 and 65 years weight gain is a major health concern. Obesity is an important risk factor for multiple diseases (e.g. metabolic syndrome, diabetes mellitus, hypertension and cardiovascular disease), and several studies have shown that the transition to menopause is associated with adverse changes in body composition. In particular, it is common to observe the accumulation of adipose tissue in the abdominal region which is believed to be an important determinant of the increase in cardiovascular risk.

The first-line strategy for weight management in overweight / obese subjects is the modification of dietary habits and lifestyle in terms of physical activity. However, nowadays, there is also a growing interest in complementary therapies (i.e. herbal supplements, acupuncture, etc ...) that can be used alone or in combination to achieve more consistent results. In this context, preliminary evidence supports the potential role of some compounds of vegetal origin such as resistant starch, epigallocatechin gallate and chlorogenic acid as adjuvants of dietary therapy for overweight.

These nutrients may be an important therapeutic aid for overweight subjects. However, in support of their use, the evidence from good quality trials is limited.

ELIGIBILITY:
Inclusion Criteria:

* menopause of recent onset
* overweight (body mass index ≥ 25) or weight gain ≥ 10% after menopause
* written informed consent

Exclusion Criteria:

* use of Orlistat
* cancer diagnosis
* unavailability to planned measurements

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Body weight | 3 months
  Difference in change in body weight between patients receiving the experimental product and those not assigned to its use

SECONDARY OUTCOMES:
Body weight | 6 months
  Difference in change in body weight between patients receiving the experimental product for 6 months and those assigned to its use for 3 months
Insulin resistance | 3 months
  Difference in change in homeostasis model assessment of insulin resistance between patients receiving the experimental product and those not assigned to its use
LDL cholesterol | 3 months
  Difference in change in LDL cholesterol between patients receiving the experimental product and those not assigned to its use
Triglycerides | 3 months
  Difference in change in triglycerides between patients receiving the experimental product and those not assigned to its use
Insulin resistance | 6 months
  Difference in change in homeostasis model assessment of insulin resistance between patients receiving the experimental product for 6 months and those assigned to its use for 3 months
LDL cholesterol | 6 months
  Difference in change in LDL cholesterol between patients receiving the experimental product for 6 months and those assigned to its use for 3 months
Triglycerides | 6 months
  Difference in change in triglycerides between patients receiving the experimental product for 6 months and those assigned to its use for 3 months
Visceral adiposity | 3 months
  Difference in change in anthropometric parameters describing fat distribution (waist circumference) between patients receiving the experimental product and those not assigned to its use
Visceral adiposity | 6 months
  Difference in change in anthropometric parameters describing fat distribution (waist circumference) between patients receiving the experimental product for 6 months and those assigned to its use for 3 months
Fat free mass | 3 months
  Difference in change in body composition parameters (measured by bioelectrical impedance analysis) between patients receiving the experimental product and those not assigned to its use
Fat free mass | 6 months
  Difference in change in body composition parameters (measured by bioelectrical impedance analysis) between patients receiving the experimental product for 6 months and those assigned to its use for 3 months
Menopausal symptoms | 3 months
  Difference in change in the severity of menopausal symptoms (using the Green Climacteric Scale) between patients receiving the experimental product and those not assigned to its use
Menopausal symptoms | 6 months
  Difference in change in the severity of menopausal symptoms (using the Green Climacteric Scale) between patients receiving the experimental product for 6 months and those assigned to its use for 3 months
Quality of life | 3 months
  Difference in change in quality of life (measured by the SF-36 Health Survey) between patients receiving the experimental product and those not assigned to its use
Quality of life | 6 months
  Difference in change in quality of life (measured by the SF-36 Health Survey) between patients receiving the experimental product for 6 months and those assigned to its use for 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Caccialanza, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Undecided